CLINICAL TRIAL: NCT06001814
Title: Mindfulness and Behavior Change to Improve Cardiovascular Health of Older People With HIV
Acronym: OM-OH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jacklyn D. Foley, Ph.D, Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023P002014; PA20-206 (Other Grant/Funding Number: NHLBI); 1K23HL167650-01A1 (NIH)
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hiv; Cardiovascular Diseases
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cardiovascular Diseases | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- One-Mind One-Heart (Experimental): One-Mind One-Heart (OM-OH) is intended to be a mindfulness-based, behavior change intervention to reduce psychological and behavioral cardiovascular disease risk.
  Interventions: Behavioral: One-Mind One-Heart
- Education (Active Comparator): The education session will provide information on behaviors important for cardiovascular disease risk reduction.
  Interventions: Other: Education

INTERVENTIONS:
Behavioral: One-Mind One-Heart — One-Mind One-Heart will include mindfulness and behavior change skills to address psychological distress, physical activity, diet, and substance use.
  Arms: One-Mind One-Heart
Other: Education — Education will be provided on behavioral cardiovascular disease risk reduction strategies, such as increasing physical activity, reducing salt intake in diet, and reduce/stop alcohol and tobacco-use.
  Arms: Education

SUMMARY:
Older people with HIV (OPWH) are disproportionately impacted by cardiovascular disease (CVD) attributable to behavioral risk factors, and chronic HIV immune dysregulation resulting inflammation. Systemic inflammation is exacerbated by psychological distress via activating the immune response and driving pro-inflammatory CVD risk behaviors. There is promising evidence to suggest that mindfulness could be an effective intervention to reduce psychological distress and support behaviorally- and inflammatory-mediated CVD risk reduction. This project aims to refine and synthesize mindfulness and behavior change content from evidence-based protocols (mindfulness-based stress reduction and diabetes prevention program) to develop and pilot test a new text message-enhanced intervention called "One Mind One Heart" (OM-OH) using feedback from semi-structured interviews with OPWH in psychological distress (N=20), and my multidisciplinary mentorship team (Aim 1). An open pilot (N=5) with exit interviews and pre-post self-report assessments, will inform the initial acceptability of OM-OH and further refine OM-OH as needed (Aim 2). Finally, a pilot randomized controlled trial (RCT; N=50) will be conducted to a.) evaluate benchmarks of feasibility and acceptability of study methods and refined OM-OH compared to enhanced usual care, and b.) investigate potential for effects on psychological distress, inflammation, and behavioral CVD risk (Aim 3). Findings will provide the foundation for an R01 application to conduct an efficacy trial of OM-OH to reduce inflammatory-mediated CVD risk among OPWH.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥50 years
2. clinical diagnosis of HIV per medical record or provision of current antiretroviral medication prescription
3. viral suppression - i.e., lower than detectable limit - per medical record or provision of viral load test from the past six months
4. current elevated psychological distress (score ≥10 on 10-item Kessler Psychological Distress Scale [K10]) screener)
5. ≥1 CVD risk factor (based on ACC/AHA Atherosclerotic Cardiovascular Disease Risk Score Calculator; e.g., diabetes, current smoker, hypertension, and high cholesterol
6. access to cell phone with text messaging capabilities

Exclusion Criteria:

1. non-English-speaking
2. cognitive impairments preventing informed consent
3. untreated or under-treated serious mental illness (i.e., psychosis and bipolar disorder) based on clinical interview

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | Baseline (pre-intervention)
  70% or more of participants consent to screening, meet screening criteria, are eligible, and agree to participate in the study
Feasibility of eligibility criteria | Baseline (pre-intervention)
  Less than 20% of participants are ineligible due to each criterion
Feasibility of randomization | Pre-intervention
  70% or more of participants are randomized and complete the first intervention session
Feasibility of the OM-OM intervention | Duration of intervention
  70% or more of participants attend all sessions and complete all homework
Feasibility of research assessments | Duration of intervention; 0 and 12-week follow-up
  70% or more of weekly and follow-up research assessments are completed
Feasibility of blood draws | Baseline; 12-week follow-up
  70% of more are collected
Acceptability of OM-OH intervention | 0-weeks post-intervention
  Rating of 7.5 or greater/10 on: session satisfaction, helpfulness, and utility; overall program satisfaction; plan to use the skills; and would recommend the intervention program to a friend
Acceptability of text-enhanced delivery | 0-weeks post-intervention
  Rating of 7.5 or greater/10 on: ease, and confidence of use; and rating of 2 or less/10 on interference of technical problems
Acceptability of blood draws | 0- and 12-weeks post-intervention
  Rating of 7.5 or greater/10 on ease of collection; and rating of 2 or less/10 on pain

SECONDARY OUTCOMES:
Five Factor Mindfulness Questionnaire (FFMQ) | 0 and 12-weeks post-intervention
  The FFQ assesses trait mindfulness.There are five sub scales: observing, describing, acting with awareness, non-judging, and non-reactivity. The FFMQ sub scale summary scores can be calculated by dividing the total in each category by the number of items in that category. The FFMQ sum score can be divided by 39 to get an average item score. Higher scores indicated greater trait mindfulness.
Patient Health Questionnaire - 9 (PHQ-9) | 0 and 12-weeks post-intervention
  PHQ-9 assesses depressive symptoms. Total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depressive symptoms, respectively.
Generalized Anxiety Disorder - 7 (GAD-7) | 0 and 12-weeks post-intervention
  GAD-7 assesses anxiety symptoms. Total scores of 5, 10, and 15 represent cut points for mild, moderate, and severe anxiety symptoms, respectively.
Perceived Stress Scale (PSS) | 0 and 12-weeks post-intervention
  The PSS assessed perceived stress. Scores on the PSS range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
HIV/AIDS Stress Scale | 0 and 12-weeks post-intervention
  The HIV/AIDS Stress Scale assesses HIV-related stress. The total score ranges from 0-68, with higher scores indicating higher levels of HIV-related stress.
Alcohol Use Disorder Identification Test - Concise (AUDIT-C) | 0 and 12-weeks post-intervention
  The AUDIT-C is scored on a scale of 0-12 (scores of 0 reflect no alcohol use). In men, a score of 4 or more is considered positive for hazardous drinking; in women, a score of 3 or more is considered positive for hazardous drinking. Generally, the higher the AUDIT-C score, the more likely it is that the patient's drinking is affecting his/her health and safety.
Physical Activity and Sedentary Behavior Questionnaire (PASBQ) | 0 and 12-weeks post-intervention
  The PASBQ assesses frequency and time spent in physical activity and sedentary behaviors. These time will be compared to Centers for Disease Control and Prevention (CDC) to determine if current guidelines are being met (yes/no) for 150 minutes of moderate aerobic activity (or 75 minutes of vigorous aerobic activity) and 2 or more days of muscle strengthening activities.
Dietary Risk Assessment (DRA) | 0 and 12-weeks post-intervention
  The DRA assesses dietary patterns. A total DRA score and 4 subscales (Nuts, Oils, Dressings, and Spreads; Vegetables, Fruit, Whole Grains, and Beans; Drinks, Desserts, Snacks, Eating Out, and Salt; and Fish, Meat, Poultry, Dairy, and Eggs) can be derived. Subscales are scored independently by assigning score values accordingly: 2 for response choices in the "Desirable" column; 1 for response choices in the "Could be improved" column; and 0 for response choices in the "Needs to be improved" column. Sum the 4 subscales to obtain a total DRA score ranging 0 to 46. For all scoring, a higher score represents a more healthful dietary pattern.
Fagerstrom Test For Nicotine Dependence (FTND) | 0 and 12-weeks post-intervention
  The FTND assesses dependence on nicotine. Scores for all item are summed. Scores of �1-2: low dependence; 3-4 low to moderate dependence; 5-7 moderate dependence; 8+ high dependence.
Inflammation Biomarkers | 0- and 12-weeks post-intervention
  Interleukin-6 and C-reactive protein measured in picograms per milliliter of blood

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
We plan to share aggregated data only.